CLINICAL TRIAL: NCT04491955
Title: Phase II Trial of Combination Immunotherapy in Subjects With Advanced Small Bowel and Colorectal Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hoyoung M. Maeng, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200138; 20-C-0138
Record Dates: First submitted 2020-07-29; First posted 2020-07-30 (Actual); Results first posted 2023-11-14 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Small Bowel Cancers; Colorectal Cancers
Keywords: CEA MUC1 Vaccine; CV301; M7824; N-803; NHS-IL12; Bintrafusp alfa; M9241
MeSH Terms: conditions — Colorectal Neoplasms | interventions — ALT-803; NHS-IL12 immunocytokine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/Arm 1 (Experimental): CEA/ MUC1 Vaccines + M7824 + N-803 (Triple Therapy).
  Interventions: Biological: CV301; Drug: MSB0011359C; Drug: N-803
- 2/Arm 2A (Experimental): CEA/ MUC1 Vaccines + M7824 + N-803 + NHSIL12 (Quadruple Therapy); dose escalation of NHS-IL12.
  Interventions: Biological: CV301; Drug: MSB0011359C; Drug: N-803; Drug: NHS-IL12
- 3/Arm 2B (Experimental): CEA/ MUC1 Vaccines + M7824 + N-803 + NHSIL12 (Quadruple Therapy); fixed dose of NHS-IL12.
  Interventions: Biological: CV301; Drug: MSB0011359C; Drug: N-803; Drug: NHS-IL12

INTERVENTIONS:
Biological: CV301 — CV301 vaccine consists of MVA-BN-CV301 and FPV-CV301. MVA-BN-CV301 (4 x 10^8 infectious units/0.5 mL each) will be administered as four subcutaneous injections on D1 and D15. Starting on D29, FPV-CV301 (1 x 10^9 infectious units/ 0.5mL) will be administered as a single subcutaneous injection every 4 weeks on Arm 1 or every 6 weeks on Arm 2A and 2B for up to one year.
Drug: MSB0011359C — Subjects will receive M7824 via IV infusion over 1 hour (-10 minutes / +20 minutes, that is, over 50 to 80 minutes) once every 2 weeks. M7824 will be administered as a "flat" dose of 1,200 mg or 300 mg independent of body weight. M7824 is administered as an intravenous infusion with a mandatory 0.2 micron in-line filter.
Drug: N-803 — N-803 will be given via subcutaneous injection at a dose of 15 mcg/kg every four weeks on Arm 1. N-803 will be administered at as dose of 10 (Micro)g/kg by SC injection every 4 weeks on Arm 2A and Arm 2B.
Drug: NHS-IL12 — NHS-IL12 will be given via subcutaneous injection at a dose of 8 mcg/kg every 4 weeks or 16 mcg/kg for the first 4 injections and 8 mcg/kg thereafter on Arms 2A and 2B.
  Arms: 2/Arm 2A; 3/Arm 2B

SUMMARY:
Background:

Metastatic or refractory/recurrent small bowel and colorectal cancers cannot be cured and are often not helped by standard treatments. Researchers want to find better treatments by testing a combination of drugs.

Objective:

To learn if a new combination of immunotherapy drugs can shrink tumors in people with advanced small bowel and colorectal cancers.

Eligibility:

People ages 18 and older who have advanced metastatic or refractory/recurrent small bowel and/or colorectal cancer.

Design:

Participants will be screened on a separate protocol. They will have a physical exam and medical history. They will have imaging scans. They will have blood and urine tests. Their heart function will be measured. They may have a tumor biopsy.

Participants will repeat some of the screening tests during the study.

Participants will be put into study groups. Each group will get a combination of the following drugs: CV301 vaccine (modified vaccinia Ankara (MVA)-BN-CV301 and Fowlpox (FPV)-CV301), M7824 (MSB0011359C), and N-803 (Anktiva). Some will also get NHS-IL12 (M9241).

Participants will get the CV301 vaccines by injection under the skin. They will get M7824 by intravenous infusion every 2 weeks. They will get N-803 by injection under the skin every 2 or 4 weeks. They may get NHS-IL12 by injection under the skin every 4 weeks. They will take the study drugs for up to 1 year. They will visit the National Institutes of Health (NIH) every 2 weeks.

After treatment ends, participants will go to the clinic for a 28-day follow-up visit or have a telephone call. They will be contacted every 3 months for 1 year, and then every 6 months after that for the rest of their life.

DETAILED DESCRIPTION:
Background:

* Metastatic or refractory/recurrent small bowel and colorectal cancers are incurable and poorly palliated by standard therapies. There is an unmet need for active treatments for these tumors.
* To date immunotherapies including anti programmed cell death protein 1 (PD-1) or anti programmed death-ligand 1 (PD-L1) inhibitors have proven largely ineffective for the vast majority of these cancers.

  * In microsatellite stable (MSS) colorectal cancer (>95% of these cancers) the response rate to checkpoint inhibitors has been <5%.
  * Preclinical studies suggest that the use of different combinations of multiple immunotherapy agents may improve anti-tumor efficacy. These studies have employed (1) a vaccine targeting a tumor associated antigen, (2) an IL-15 superagonist (N-803, also known as ALT-803), (3) an anti-PD-L1 MAb or a bifunctional fusion protein targeting PD-L1 and TGF beta (M7824 (MSB0011359C), and (4) a tumor targeted immunocytokine (NHS-IL12 (M9241).

Objectives:

To evaluate the objective response rate (ORR) according to Response Evaluation Criteria (Response Evaluation Criteria in Solid Tumors (RECIST) 1.1) of the combination of (1) CV301, a poxviral based vaccine targeting carcinoembryonic antigen (CEA) and mucin-1 (MUC1), (2) N-803 and (3) M7824; and of the combination of (1) CV301, (2) N-803, (3) M7824 and (4) NHS-IL12 (M9241) in subjects with advanced checkpoint naive microsatellite stable (MSS) small bowel and colorectal cancers.

Eligibility:

* Age >= 18 years old
* Subjects with cytologically or histologically confirmed locally advanced or metastatic small bowel or colorectal adenocarcinomas.
* Prior first line systemic therapy is required unless the patient declines standard treatment after appropriate counseling has been provided.
* Subjects must have measurable disease.

Design:

* This is a phase II trial of combination immunotherapy, with a brief dose escalation portion for Arm 2.
* The trial will be conducted using a Simon optimal two-stage design in each Phase II Arm.
* Patients will be enrolled on the following arms in sequential order: (1) Arm 1: CV301 + M7824 + N-803, (2) Arm 2A and Arm 2B: CV301 + M7824 + N-803 + NHS-IL12; N-803 dose level will be evaluated in Arm 2A prior to further enrollment in Arm 2B.
* The first six patients on arm 1 will be evaluable for dose limiting toxicities (DLTs) and accrual will only continue to 9 patients on that arm if less than 2 out of the first 6 patients experience a DLT.
* In Arm 2B, patients will receive 4 drug treatments (CV301 + M7824 + N-803 + NHSIL12), but the dose level of N-803 will first be determined during a 3-level dose escalation portion, Arm 2A. Following determination of the maximum tolerated dose (MTD) or highest safe dose evaluated, the 6 patients at that dose level will be included among the initial 9 patients for the first stage of that arm.
* If two or more out of nine patients have objective responses on a given arm that arm will be expanded to enroll 20 evaluable patients.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Subjects with cytologically or histologically confirmed locally advanced or metastatic small bowel or colorectal adenocarcinoma
2. Subjects must have received two prior lines of systemic therapy unless the subject is not eligible to receive standard therapy or declines standard treatment
3. Subjects must have measurable disease
4. Eastern Cooperative Oncology Group (ECOG) performance status <= 2
5. Adequate hematologic function at screening, as follows:

   * Absolute neutrophil count (ANC) >=1 x 10^9/L
   * Hemoglobin >= 9 g/dL
   * Platelets >= 75,000/microliter
6. Adequate renal and hepatic function at screening, as follows:

   - Serum creatinine <= 1.5 x upper limit of normal (ULN) OR

   Measured or calculated creatinine clearance >= 40 mL/min for participant with creatinine levels > 1.5 X institutional ULN (glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl);
   * Bilirubin <= 1.5 x ULN OR in subjects with Gilbert's syndrome, a total bilirubin <= 3.0 x ULN
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 2.5 x ULN, unless liver metastases are present, then values must be <= 3 x ULN)
7. The effects of the immunotherapies on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study treatment and up to two months after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
8. Participants serologically positive for human immunodeficiency virus (HIV), Hep B, Hep C are eligible as long as the viral loads are undetectable by quantitative polymerase chain reaction (PCR). HIV positive participants must have cluster of differentiation 4 (CD4) count >= 200 cells per cubic millimeter at enrollment, be on stable antiretroviral therapy for at least 4 weeks and have no reported opportunistic infections or Castleman s disease within 12 months prior to enrollment.
9. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Participants with prior investigational drug, chemotherapy, immunotherapy or any prior radiotherapy (except for palliative bone directed therapy) within the past 28 days prior to the first drug administration except if the investigator has assessed that all residual treatment-related toxicities have resolved or are minimal and feel the participant is otherwise suitable for enrollment. Additionally, current therapies (e.g., maintenance capecitabine) may be continued where in the opinion of the investigator stopping such therapies may increase the risk of disease progression. Also, participants may continue adjuvant hormonal therapy in the setting of a definitively treated cancer (e.g., breast).
2. Participants with microsatellite unstable or mismatch repair deficient disease.
3. Major surgery within 28 days prior to the first drug administration (minimally invasive procedures such as diagnostic biopsies are permitted).
4. Known life-threatening side effects resulting from prior checkpoint inhibitor therapy (e.g., colitis, pneumonitis, fulminant hepatitis which led to permanent discontinuation of prior checkpoint therapy). Autoimmune toxicity which was not life threatening (e.g., arthritis) or did not lead to discontinuation of prior checkpoint therapy is allowed.
5. Known active brain or central nervous system metastasis (less than a month out from definitive radiotherapy or surgery), seizures requiring anticonvulsant treatment (<3 months) or clinically significant cerebrovascular accident (<3 months). In order to be eligible participants must have repeat central nervous system (CNS) imaging at least a month after definitive treatment showing stable CNS disease. Participants with evidence of intra-tumoral or peritumoral hemorrhage on baseline imaging are also excluded unless the hemorrhage is grade <= 1 and has been shown to be stable on two consecutive imaging scans.
6. Pregnant women are excluded from this study because these drugs have not been tested in pregnant women and there is potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these immunotherapies, breastfeeding should be discontinued if the mother is treated on this protocol.
7. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent with exception of:

   * Diabetes type I, eczema, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease or other mild autoimmune disorders not requiring immunosuppressive treatment;
   * Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses <= 10 mg of prednisone or equivalent per day;
   * Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable;
   * Subjects on systemic intravenous or oral corticosteroid therapy with the exception of physiologic doses of corticosteroids (<= the equivalent of prednisone 10 mg/day) or other immunosuppressive agents such as azathioprine or cyclosporin A are excluded on the basis of potential immune suppression. For these subjects these excluded treatments must be discontinued at least 1 weeks prior to enrollment for recent short course use (<= 14 days) or discontinued at least 4 weeks prior to enrollment for long term use (> 14 days). In addition, the use of corticosteroids as premedication for contrast-enhanced studies is allowed prior to enrollment and on study.
8. Subjects with a history of serious intercurrent chronic or acute illness, such as cardiac or pulmonary disease, hepatic disease, bleeding diathesis or recent (within 3 months) clinically significant bleeding events or other illness considered by the Investigator as high risk for investigational drug treatment.
9. Subjects unwilling to accept blood products as medically indicated.
10. History of second malignancy within 3 years of enrollment except for the following: adequately treated localized skin cancer, cervical carcinoma in situ, superficial bladder cancer, or other localized malignancy which has been adequately treated or malignancy which does not require active systemic treatment (e.g., low risk chronic lymphocytic leukemia (CLL).
11. Subjects with a known severe hypersensitivity reaction to a monoclonal antibody (grade >= 3 National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE v5) will be evaluated by the allergy/immunology team prior to enrollment.
12. Receipt of any organ transplantation requiring ongoing immunosuppression.
13. Receipt of prior lymphodepleting chemotherapy (e.g., cyclophosphamide or fludarabine at standard lymphodepleting doses).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2024-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hoyoung Maeng, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the Database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the Database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Bracken-Clarke D, Pastor DM, Marte JL, Donahue RN, Hodge JW, Cordes L, Floudas CS, Tschernia NP, Karzai F, Brownell I, Turkbey EB, Soon-Shiong P, Schlom J, Gulley JL, Maeng HM, Strauss J, Redman JM. The Quadruple Immunotherapy for Colorectal Cancer (QuICC) Trial for Mismatch Repair-Proficient Metastatic Colorectal Cancer. Oncologist. 2026 Jan 10:oyag008. doi: 10.1093/oncolo/oyag008. Online ahead of print. PMID 41520164
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0138.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1, Arm 1 Triple Therapy Without NHS-IL12 (M9241): Carcinoembryonic antigen (CEA)/ Mucin 1 (MUC1) Vaccines + (M7824 (MSB0011359C) + N-803 (Anktiva) (Triple Therapy).
  CV301: CV301 vaccine consists of modified vaccinia Ankara (MVA)-BN-CV301 and Fowlpox (FPV)-CV301). MVA-BN-CV301 (4 x 10^8 infectious units/0.5 mL each) will be administered as four subcutaneous (SC) injections on Day (D)1 and D15. Starting on D29, FPV-CV301 (1 x 10^9 infectious units/ 0.5mL) will be administered as a single subcutaneous injection every 4 weeks on Arm 1 or every 6 weeks on Arm 2A and 2B for up to one year.
  MSB0011359C: Participants will receive M7824 via intravenous (IV) infusion over 1 hour (-10 minutes / +20 minutes, that is, over 50 to 80 minutes) once every 2 weeks. M7824 will be administered as a "flat" dose of 1,200 mg or 300 mg independent of body weight. M7824 is administered as an intravenous infusion with a mandatory 0.2 micron in-line filter.
  N-803: N-803 will be given via subcutaneous injection at a dose of 15 mcg/kg every four weeks on Arm 1. N-803 will be administered at as dose of 10 (Micro)g/kg by SC injection every 4 weeks on Arm 2A and Arm 2B.
- Cohort 2, Arm 2a Dose Level (DL) 1, Quad Therapy Dose Escalation: Carcinoembryonic antigen (CEA)/ Mucin 1 (MUC1) Vaccines + M7824 (MSB0011359C) + N-803 (Anktiva) + (NHS-IL12 (M9241) (Quadruple Therapy); dose escalation of NHS-IL12.
  CV301: CV301 vaccine consists of modified vaccinia Ankara (MVA)-BN-CV301 and Fowlpox (FPV)-CV301). MVA-BN-CV301 (4 x 10^8 infectious units/0.5 mL each) will be administered as four subcutaneous (SC) injections on Day (D1) and D15. Starting on D29, FPV-CV301 (1 x 10^9 infectious units/ 0.5mL) will be administered as a single subcutaneous injection every 4 weeks on Arm 1 or every 6 weeks on Arm 2A and 2B for up to one year.
  MSB0011359C: Participants will receive M7824 via intravenous (IV) infusion over 1 hour (-10 minutes / +20 minutes, that is, over 50 to 80 minutes) once every 2 weeks. M7824 will be administered as a "flat" dose of 1,200 mg or 300 mg independent of body weight. M7824 is administered as an intravenous infusion with a mandatory 0.2 micron in-line filter.
  N-803: N-803 will be given via subcutaneous injection at a dose of 15 mcg/kg every four weeks on Arm 1. N-803 will be administered at as dose of 10 (Micro)g/kg by SC injection every 4 weeks on Arm 2A and Arm 2B.
  NHS-IL12: NHS-IL12 will be given via subcutaneous injection at a dose of 8 mcg/kg every 4 weeks or 16 mcg/kg for the first 4 injections and 8 mcg/kg thereafter on Arms 2A and 2B.
- Cohort 2, Arm 2a, Dose Level (DL) DL2, Quad Therapy Dose Escalation: Carcinoembryonic antigen (CEA)/Mucin-1 (MUC-1) Vaccines + M7824 (MSB0011359C) + N-803 (Anktiva) + NHS-IL12 (M9241) (Quadruple Therapy); dose escalation of NHS-IL12.
  CV301: CV301 vaccine consists of modified vaccinia Ankara (MVA)-BN-CV301 and FPV-CV301. MVA-BN-CV301 (4 x 10^8 infectious units/0.5 mL each) will be administered as four subcutaneous (SC) injections on Day (D)1 and D15. Starting on D29, FPV-CV301 (1 x 10^9 infectious units/ 0.5mL) will be administered as a single subcutaneous injection every 4 weeks on Arm 1 or every 6 weeks on Arm 2A and 2B for up to one year.
  MSB0011359C: Participants will receive M7824 via intravenous (IV) infusion over 1 hour (-10 minutes / +20 minutes, that is, over 50 to 80 minutes) once every 2 weeks. M7824 will be administered as a "flat" dose of 1,200 mg or 300 mg independent of body weight. M7824 is administered as an intravenous infusion with a mandatory 0.2 micron in-line filter.
  N-803: N-803 will be given via subcutaneous injection at a dose of 15 mcg/kg every four weeks on Arm 1. N-803 will be administered at as dose of 10 (Micro)g/kg by SC injection every 4 weeks on Arm 2A and Arm 2B.
  NHS-IL12: NHS-IL12 will be given via subcutaneous injection at a dose of 8 mcg/kg every 4 weeks or 16 mcg/kg for the first 4 injections and 8 mcg/kg thereafter on Arms 2A and 2B.
- Cohort 2, Arm 2b Dose Level (DL)2, Quad Therapy Fixed Dose: Carcinoembryonic antigen (CEA)/Mucin-1 (MUC-1) Vaccines + M7824 (MSB0011359C) + N-803 (Anktiva) + NHS-IL12 (M9241) (Quadruple Therapy); fixed dose of NHS-IL12.
  CV301: CV301 vaccine consists of modified vaccinia Ankara (MVA)-BN-CV301 and Fowlpox (FPV)-CV301). MVA-BN-CV301 (4 x 10^8 infectious units/0.5 mL each) will be administered as four subcutaneous (SC) injections on Day (D)1 and D15. Starting on D29, FPV-CV301 (1 x 10^9 infectious units/ 0.5mL) will be administered as a single subcutaneous injection every 4 weeks on Arm 1 or every 6 weeks on Arm 2A and 2B for up to one year.
  MSB0011359C: Participants will receive M7824 via intravenous (IV) infusion over 1 hour (-10 minutes / +20 minutes, that is, over 50 to 80 minutes) once every 2 weeks. M7824 will be administered as a "flat" dose of 1,200 mg or 300 mg independent of body weight. M7824 is administered as an intravenous infusion with a mandatory 0.2 micron in-line filter.
  N-803: N-803 will be given via subcutaneous injection at a dose of 15 mcg/kg every four weeks on Arm 1. N-803 will be administered at as dose of 10 (Micro)g/kg by SC injection every 4 weeks on Arm 2A and Arm 2B.
  NHS-IL12: NHS-IL12 will be given via subcutaneous injection at a dose of 8 mcg/kg every 4 weeks or 16 mcg/kg for the first 4 injections and 8 mcg/kg thereafter on Arms 2A and 2B.
Period: Overall Study
Arm/Group | Cohort 1, Arm 1 Triple Therapy Without NHS-IL12 (M9241) | Cohort 2, Arm 2a Dose Level (DL) 1, Quad Therapy Dose Escalation | Cohort 2, Arm 2a, Dose Level (DL) DL2, Quad Therapy Dose Escalation | Cohort 2, Arm 2b Dose Level (DL)2, Quad Therapy Fixed Dose
Started | 12 | 8 | 6 | 6
Completed | 12 | 8 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Arm 1 Triple Therapy Without NHS-IL12 (M9241) | Cohort 2, Arm 2a Dose Level (DL) 1, Quad Therapy Dose Escalation | Cohort 2, Arm 2a, Dose Level (DL) DL2, Quad Therapy Dose Escalation | Cohort 2, Arm 2b Dose Level (DL)2, Quad Therapy Fixed Dose | Total
Number analyzed (Participants) | 12 | 8 | 6 | 6 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 6 | 4 | 5 | 26
  >=65 years | 1 | 2 | 2 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.27 (8.31) | 56.64 (13.82) | 50.72 (16.47) | 58.85 (5.7) | 55.43 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 1 | 4 | 17
  Male | 4 | 4 | 5 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 8 | 6 | 6 | 31
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 0 | 0 | 5
  White | 6 | 6 | 6 | 5 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 6 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) for Triple Therapy
Description: ORR of the combination of (1) Carcinoembryonic antigen (CEA)/Mucin-1 (MUC1) vaccines, (2) N-803 (Anktiva) and (3) M7824 (MSB0011359C) in participants with advanced small bowel and colorectal cancers was evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Objective response is a complete or partial radiographic response as defined by RECIST 1.1. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: one year
Measure: Number; unit: Proportion of participants
Arm/Group | Cohort 1, Arm 1 Triple Therapy Without NHS-IL12 (M9241)
Number analyzed (Participants) | 12
Proportion of participants
  Complete Response | 0
  Partial Response | 0

2. Primary Outcome: Objective Response Rate (ORR) for Quadruple Therapy
Description: ORR of the combination of (1) Carcinoembryonic antigen (CEA)/Mucin-1 (MUC1) vaccines, (2) N-803 (Anktiva), (3) M7824 (MSB0011359C) and (4) NHS-IL12 (M9241) in participants with advanced small bowel and colorectal cancers was evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Objective response is a complete or partial radiographic response as defined by RECIST 1.1. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: one year
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 2, Arm 2a Dose Level (DL) 1, Quad Therapy Dose Escalation | Cohort 2, Arm 2a, Dose Level (DL) DL2, Quad Therapy Dose Escalation | Cohort 2, Arm 2b Dose Level (DL)2, Quad Therapy Fixed Dose
Number analyzed (Participants) | 8 | 6 | 6
Percentage of participants
  Complete Response | 12.5 | 0 | 0
  Partial Response | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Grade 3, Grade 4, and/or Grade 5 Adverse Events Related to Triple Therapy
Description: Safety of the combination of (1) CV301, (2) N-803 (Anktiva) and (3) M7824 (MSB0011359C) in participants with advanced small bowel and colorectal cancers was assessed using the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to date off study, approximately 29 months and 1 day for Cohort 1, Arm 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Arm 1 Triple Therapy Without NHS-IL12 (M9241)
Number analyzed (Participants) | 12
Participants
  Grade 3 Alkaline phosphatase increased | 1
  Grade 3 Anemia | 1
  Grade 3 Aspartate aminotransferase increased | 1
  Grade 3 Cardiac troponin I increased | 1
  Grade 4 | 0
  Grade 5 | 0

4. Secondary Outcome: Number of Participants With Grade 3, Grade 4, and/or Grade 5 Adverse Events Related to Quadruple Therapy
Description: Safety of the combination of (1) CV301, (2) N-803 (Anktiva), (3) M7824 (MSB0011359C) and (4) NHS-IL12 (M9241) in participants with advanced small bowel and colorectal cancers was assessed using the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to date off study, approximately 27 months for Cohort 2, Arm 2a Dose Level 1; 18 months and 29 days for cohort 2, Arm 2a Dose Level 2; and 7 months and 20 days for Cohort 2, Arm 2b, Dose Level 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2, Arm 2a Dose Level (DL) 1, Quad Therapy Dose Escalation | Cohort 2, Arm 2a, Dose Level (DL) DL2, Quad Therapy Dose Escalation | Cohort 2, Arm 2b Dose Level (DL)2, Quad Therapy Fixed Dose
Number analyzed (Participants) | 8 | 6 | 6
Participants
  Grade 3 Anemia | 3 | 1 | 0
  Grade 3 Duodenal hemorrhage | 1 | 0 | 0
  Grade 3 Adrenal insufficiency | 0 | 1 | 0
  Grade 3 General disorders & administration site conditions - Mucosal bleeding, lower GI hemorrhage | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS per treatment assignment (three or four drug combination was evaluated using Kaplan-Meier methods and is defined as the time from the date of first treatment to the date of disease progression or death (any cause) whichever occurs first. Participants who do not have disease progression or have not died at the end of follow up will be censored at the last known date the participant was progression free. Progression was assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and is defined as the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: From time to enrollment up to 35 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1, Arm 1 Triple Therapy Without NHS-IL12 (M9241) | Cohort 2, Arm 2a Dose Level (DL) 1, Quad Therapy Dose Escalation | Cohort 2, Arm 2a, Dose Level (DL) DL2, Quad Therapy Dose Escalation | Cohort 2, Arm 2b Dose Level (DL)2, Quad Therapy Fixed Dose
Number analyzed (Participants) | 12 | 8 | 6 | 6
Months | 1.8 [1.8 to NA] — The confidence intervals are calculated using the Brookmeyer-Crowley method; if the upper limit of the interval does not intersect the median then it is not able to be estimated. | 1.8 [1.8 to NA] — The confidence intervals are calculated using the Brookmeyer-Crowley method; if the upper limit of the interval does not intersect the median then it is not able to be estimated. | 1.8 [1.8 to NA] — The confidence intervals are calculated using the Brookmeyer-Crowley method; if the upper limit of the interval does not intersect the median then it is not able to be estimated. | 0.92 [0.92 to NA] — The confidence intervals are calculated using the Brookmeyer-Crowley method; if the upper limit of the interval does not intersect the median then it is not able to be estimated.

6. Secondary Outcome: Overall Survival (OS)
Description: OS per treatment assignment (three or four drug combination) evaluated using Kaplan-Meier methods. OS is defined as the time from the date of first treatment to the date of death (any cause). Participants who are alive at the end of follow up will be censored at the last known date alive.
Time Frame: Up to 35 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1, Arm 1 Triple Therapy Without NHS-IL12 (M9241) | Cohort 2, Arm 2a Dose Level (DL) 1, Quad Therapy Dose Escalation | Cohort 2, Arm 2a, Dose Level (DL) DL2, Quad Therapy Dose Escalation | Cohort 2, Arm 2b Dose Level (DL)2, Quad Therapy Fixed Dose
Number analyzed (Participants) | 12 | 8 | 6 | 6
Months | 19 [12 to NA] — The confidence intervals are calculated using the Brookmeyer-Crowley method; if the upper limit of the interval does not intersect the median then it is not able to be estimated. | 19 [15 to NA] — The confidence intervals are calculated using the Brookmeyer-Crowley method; if the upper limit of the interval does not intersect the median then it is not able to be estimated. | 4.5 [4.5 to NA] — The confidence intervals are calculated using the Brookmeyer-Crowley method; if the upper limit of the interval does not intersect the median then it is not able to be estimated. | 7.0 [4.9 to NA] — The confidence intervals are calculated using the Brookmeyer-Crowley method; if the upper limit of the interval does not intersect the median then it is not able to be estimated.

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR per treatment assignment (three or four drug combination) is measured from the time measurement criteria are met for Complete Response (CR) or Partial Response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR is disappearance of all target lesions. PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 34 months
Population: 1/32 participants were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1, Arm 1 Triple Therapy Without NHS-IL12 (M9241) | Cohort 2, Arm 2a Dose Level (DL) 1, Quad Therapy Dose Escalation | Cohort 2, Arm 2a, Dose Level (DL) DL2, Quad Therapy Dose Escalation | Cohort 2, Arm 2b Dose Level (DL)2, Quad Therapy Fixed Dose
Number analyzed (Participants) | 0 | 1 | 0 | 0
Months |  | 34 [NA to NA] — 95% confidence interval cannot be calculated for one participant. |  |

8. Secondary Outcome: Number of Participants Hospitalized Due to Serious Adverse Events Attributed to Progressive Disease (PD)
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. And progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is defined as appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: time participant is first enrolled to time participant is taken off of study treatment, an average of 2.1 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Arm 1 Triple Therapy Without NHS-IL12 (M9241) | Cohort 2, Arm 2a Dose Level (DL) 1, Quad Therapy Dose Escalation | Cohort 2, Arm 2a, Dose Level (DL) DL2, Quad Therapy Dose Escalation | Cohort 2, Arm 2b Dose Level (DL)2, Quad Therapy Fixed Dose
Number analyzed (Participants) | 12 | 8 | 6 | 6
Participants | 1 | 1 | 0 | 0

9. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 29 months and 1 day for Cohort 1, Arm 1; 27 months for Cohort 2, Arm 2a Dose Level (DL) 1; 18 months and 29 days for cohort 2, Arm 2a DL 2; and 7 months and 20 days for Cohort 2, Arm 2b, DL 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Arm 1 Triple Therapy Without NHS-IL12 (M9241) | Cohort 2, Arm 2a Dose Level (DL) 1, Quad Therapy Dose Escalation | Cohort 2, Arm 2a, Dose Level (DL) DL2, Quad Therapy Dose Escalation | Cohort 2, Arm 2b Dose Level (DL)2, Quad Therapy Fixed Dose
Number analyzed (Participants) | 12 | 8 | 6 | 6
Participants | 12 | 8 | 6 | 6

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 29 months and 1 day for Cohort 1, Arm 1; 27 months for Cohort 2, Arm 2a Dose Level (DL) 1; 18 months and 29 days for cohort 2, Arm 2a DL 2; and 7 months and 20 days for Cohort 2, Arm 2b, DL 2.
Arm/Group | Cohort 1, Arm 1 Triple Therapy Without NHS-IL12 (M9241) | Cohort 2, Arm 2a Dose Level (DL) 1, Quad Therapy Dose Escalation | Cohort 2, Arm 2a, Dose Level (DL) DL2, Quad Therapy Dose Escalation | Cohort 2, Arm 2b Dose Level (DL)2, Quad Therapy Fixed Dose
All-Cause Mortality (participants affected / at risk) | 9/12 | 5/8 | 4/6 | 3/6
Serious Adverse Events (participants affected / at risk) | 2/12 | 4/8 | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 12/12 | 8/8 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Arm 1 Triple Therapy Without NHS-IL12 (M9241) (N=12) | Cohort 2, Arm 2a Dose Level (DL) 1, Quad Therapy Dose Escalation (N=8) | Cohort 2, Arm 2a, Dose Level (DL) DL2, Quad Therapy Dose Escalation (N=6) | Cohort 2, Arm 2b Dose Level (DL)2, Quad Therapy Fixed Dose (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Mucosal bleeding, Lower Gastrointestinal Hemorrhage
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Arm 1 Triple Therapy Without NHS-IL12 (M9241) (N=12) | Cohort 2, Arm 2a Dose Level (DL) 1, Quad Therapy Dose Escalation (N=8) | Cohort 2, Arm 2a, Dose Level (DL) DL2, Quad Therapy Dose Escalation (N=6) | Cohort 2, Arm 2b Dose Level (DL)2, Quad Therapy Fixed Dose (N=6)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 1 (1) | 3 (4) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (5) | 2 (3) | 3 (3) | 0 (0)
Alkaline phosphatase increased (Investigations) | 3 (7) | 1 (1) | 1 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (10) | 7 (19) | 4 (4) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 4 (5) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (7) | 5 (10) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (2)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (3) | 1 (1) | 1 (2) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (4)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (3) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, conjunctival hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 3 (4) | 5 (7) | 3 (4)
Fever (General disorders) | 4 (5) | 1 (1) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 11 (20) | 7 (22) | 6 (15) | 6 (15)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Epistaxis, nose bleeding (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, MUCOSAL BLEEDING (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mucosal bleeding, epistaxis - intermittent
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mucosal bleeding, oral hemorrhage - intermittent when brushing teeth; expected
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mucosal bleeding, oral hemorrhage; mild bleeding when brushing teeth
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mucosal bleeding, epistaxis intermittent - blood tinge when blowing nose
General disorders and administration site conditions - Other, Mucosal bleeding (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mucosal bleeding, hemorrhoidal hemorrhage
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mucosal bleeding, nasopharyneal/post-nasal hemorrhage
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mucosal bleeding, oral hemorrhage - mild bleeding when brushing teeth
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mucosal bleeding, oral hemorrhage intermittent when brushing teeth
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mucosal bleeding intermittent when blows nose
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Other: mucosal bleeding, expected; epistaxis, intermittent, mild
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Vaccination site lymphadenopathy, left groin lump
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — mucosal bleeding, oral hemorrhage: mild bleeding when brushing teeth
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Hematuria (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 12 (29) | 8 (16) | 4 (17) | 6 (15)
Injury, poisoning and procedural complications - Other, Left 2nd toe wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (5) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (3) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, KERATOSIS PILARIS, bilateral arms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Weight loss (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT04491955/Prot_SAP_003.pdf
  • Informed Consent Form (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT04491955/ICF_001.pdf